CLINICAL TRIAL: NCT03161613
Title: Postmarketing Study to Assess the Safety of Nivolumab as a First- and Second-line Treatment in Patients With Metastatic Melanoma or as a Second-line Treatment for Metastatic Lung Cancer (Squamous and Nonsquamous), Metastatic Renal Cancer, Squamous Cell Carcinoma of the Head and Neck, and Chronic Hodgkin Lymphoma in Adult Patients in Mexico
Brief Title: Study to Assess the Safety of Nivolumab in the Treatment of Metastatic Melanoma, Lung Cancer, Renal Cancer, Squamous Cell Carcinoma of the Head and Neck, and Chronic Hodgkin Lymphoma in Adults in Mexico
Status: Withdrawn | Type: Observational
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-869
Record Dates: First submitted 2017-05-18; First posted 2017-05-22 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Multiple Indications Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cancer patients in Mexico: lung cancer, melanoma cancer, renal cancer, Squamous Cell Carcinoma of the Head and Neck, and chronic Hodgkin Lymphoma patients in Mexico who have failed at least one treatment before being treated with nivolumab
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
This is a post-marketing study of patients who started nivolumab as first- or second-line therapy for metastatic melanoma or as second-line therapy for metastatic squamous non-small cell lung cancer (SqNSCLC) , metastatic non-SqNSCLC, metastatic renal cell carcimona (RCC), or recurrent or metastatic squamous cell carcinoma of the head and neck cancer (SCCHN), or third-line therapy for classical Hodgkin lymphoma (cHL) in Mexico.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adult patients > 18 years of age who have a confirmed diagnosis of advanced or metastatic melanoma and is indicated for the treatment of advanced (unresectable or metastatic) melanoma; metastatic NSCLC; metastatic RCC; recurrent or metastatic SCCHN; or cHL in Mexico
2. Male and female adult patients > 18 years of age who completed the following lines of therapy: first-line platinum treatment for metastatic SqNSCLC or non-SqNSCLC; 1 first-line treatment for metastatic RCC; first-line platinum therapy for SCCHN; or bretuximab vedontin for the treatment of cHL
3. Patients who present with brain metastases are allowed, if asymptomatic, do not have edema, and are not receiving corticosteroids or radiation
4. Patients have received at least 1 dose of nivolumab

Exclusion Criteria:

1. The exclusion criteria are at the discretion of the physician. The physician should use his or her clinical judgement and international recommendations when determining eligibility. The patient will be excluded if he or she does not want to start or continue treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who started nivolumab as first- or second-line therapy for metastatic melanoma or as second-line therapy for metastatic squamous non-small cell lung cancer (SqNSCLC) , metastatic non-SqNSCLC, metastatic renal cell carcimona (RCC), or recurrent or metastatic squamous cell carcinoma of the head and neck cancer (SCCHN), or third-line therapy for classical Hodgkin lymphoma (cHL) in Mexico.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of subjects who report on-study Adverse Events(AEs) | approximately 24 months
incidence of subjects who report on-study Serious Adverse Events(SAEs) | approximately 24 months

SECONDARY OUTCOMES:
Distribution of on-study AEs | approximately 24 months
Distribution of on-study SAEs | approximately 24 months
Distribution of drug-related AEs | approximately 24 months
Distribution of drug-related SAEs | approximately 24 months
Distribution of AEs leading to discontinuation | approximately 24 months
Distribution of SAEs leading to discontinuation | approximately 24 months
Distribution of age in patients | At Baseline
Distribution of gender in patients | At Baseline
Distribution of tumor history in patients | At Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Mexico City, Mexico City, Mexico

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm